CLINICAL TRIAL: NCT05031559
Title: Episodic Future Thinking and Compassion Reduce Public Health Guideline Noncompliance Urges: A Randomised Controlled Trial
Brief Title: Episodic Future Thinking and Compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Martin & Loreto Hosking's Three Springs Foundation (Unknown); Australian Research Council (Unknown)
Responsible Party: Principal Investigator, Antonio Verdejo-García, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 26253
Record Dates: First submitted 2021-08-23; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Compliant Behavior; Self-Control; Impulsive Behavior
Keywords: Episodic future thinking; Compassion; Impulsivity; Self-control; Pandemic; Public Health
MeSH Terms: conditions — Cooperative Behavior; Self-Control; Impulsive Behavior | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not made aware whether they were in the control group or in one of the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Episodic Future Thinking (Experimental)
  Interventions: Behavioral: Episodic Future Thinking
- Compassion (Experimental)
  Interventions: Behavioral: Compassion Training
- Control (Sham Comparator)
  Interventions: Behavioral: Sham

INTERVENTIONS:
Behavioral: Episodic Future Thinking — Participants are invited to imagine themselves in a positive situation after COVID-19 public health restrictions and guidelines are lifted. They are then reminded that their actions are able to change how soon this future can be achieved.
  Arms: Episodic Future Thinking
Behavioral: Compassion Training — Participants are invited to imagine themselves in someone else's situation, who is in a bad situation due to COVID-19 (e.g., ER nurse, family of someone in ICU). They are then reminded that their decisions have an impact on the occurrence of these situations.
  Arms: Compassion
Behavioral: Sham — Participants are invited to reflect on some COVID-19 related news, and reminded that their actions have bearing on the COVID-19 situation.
  Arms: Control

SUMMARY:
During the COVID-19 (Coronavirus Disease 2019) pandemic, public health departments have issued guidelines to limit viral transmission. In this environment, people will feel urges to engage in activities that violate these guidelines, but research on guideline adherence has been reliant on surveys asking people to self-report their typical behaviour, which may fail to capture these urges as they unfold. Guideline adherence could be improved through behaviour change interventions, but considering the wide range of behaviours that COVID-19 guidelines prescribe, there are few methods that allow observing changes of aggregate guideline adherence in the 'wild'. In order to administer interventions and to obtain contemporaneous data on a wide range of behaviours, the researchers use ecological momentary assessment. In this preregistered parallel randomised trial, 95 participants aged 18-65 from the United Kingdom were assigned to three conditions using blinded block randomisation, and engage in episodic future thinking (n = 33), compassion exercises (n = 31), or a sham procedure (n = 31) and report regularly on the intensity of their occurrent urges (min. 1, max. 10) and their ability to control them. The researchers investigate whether state impulsivity and vaccine attitudes predict guideline adherence, while assessing through which mechanism these predictors affect behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Resides in the United Kingdom
* Fluent in English
* Must pass attention check in eligibility survey

Exclusion Criteria:

* Less than 50% compliance with ecological momentary assessment surveys

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-04-04 (Actual)

PRIMARY OUTCOMES:
Average strength of urges in ecological momentary assessment surveys | Multiple times per day, for one week.
  Throughout each day, participants would receive 5 ecological momentary assessment surveys that were available for 1 hour. In randomised order, they were asked whether since the last survey they had felt an urge to not wash their hands, not cover their mouths when coughing or sneezing, not socially distance (e.g. to hug, shake hands), not leave details for contact tracing, or whether they had felt an urge to leave their house, touch their face, or avoid getting tested when it would have been better to do the opposite - from a COVID-19 standpoint. Participants responded using a slider [0,10], where 0 indicated no urge, 1 indicated a very weak urge, and 10 indicated a very strong urge.
Average probability of controlling urges in ecological momentary assessment surveys | Multiple times per day, for one week.
  Throughout each day, participants would receive 5 ecological momentary assessment surveys that were available for 1 hour. In randomised order, they were asked whether since the last survey they had felt an urge to not wash their hands, not cover their mouths when coughing or sneezing, not socially distance (e.g. to hug, shake hands), not leave details for contact tracing, or whether they had felt an urge to leave their house, touch their face, or avoid getting tested when it would have been better to do the opposite - from a COVID-19 standpoint. Participants responded using a slider [0,10], where 0 indicated no urge, 1 indicated a very weak urge, and 10 indicated a very strong urge. Following that urge, participants are asked whether they gave in to that urge.

SECONDARY OUTCOMES:
Average number of resisted urges | Multiple times per day, for one week.
  Throughout each day, participants would receive 5 ecological momentary assessment surveys that were available for 1 hour. In randomised order, they were asked whether since the last survey they had felt an urge to not wash their hands, not cover their mouths when coughing or sneezing, not socially distance (e.g. to hug, shake hands), not leave details for contact tracing, or whether they had felt an urge to leave their house, touch their face, or avoid getting tested when it would have been better to do the opposite - from a COVID-19 standpoint. Participants responded using a slider [0,10], where 0 indicated no urge, 1 indicated a very weak urge, and 10 indicated a very strong urge. Following that urge, participants are asked whether they tried to resist that urge.

CONTACTS AND LOCATIONS:
Locations (1):
- Prolific online participant recruitment platform, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data are available on the Open Science Foundation (OSF) website.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data are permanently available.
URL: https://osf.io/5duvx/?view_only=d360db6dd6064aba99ec47b943adf94e